CLINICAL TRIAL: NCT00158249
Title: Cannabis Dependence: Imaging and Medication Development - 1
Brief Title: Effects of Citicoline on Brain Function and Behavior in Marijuana-Dependent Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Scott Lukas, Director, MIC & BPRL, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-19238-1; R01DA019238 (NIH); DPMC (Other: NIDA); R01DA024007 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Marijuana Abuse
Keywords: citicoline, drug abuse, marijuana
MeSH Terms: conditions — Marijuana Abuse; Substance-Related Disorders | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): matched capsules
  Interventions: Drug: placebo
- citicoline (Experimental): 2 gm/day
  Interventions: Drug: citicoline

INTERVENTIONS:
Drug: citicoline — 2 gm/day, 8 weeks treatment
  Arms: citicoline
Drug: placebo — matched for physical appearance
  Arms: placebo

SUMMARY:
The Three Aims of this study are (only studies for Aim 1 were completed)

1. Measure the impact of citicoline on marihuana use patterns in subjects' individualized natural settings and responses to marihuana challenge using functional brain MRI scans.

   Hypothesis - 2 g/day citicoline will produce greater reductions in marihuana use and craving in heavy marihuana users than placebo citicoline over a 8-week treatment period as measured in their natural environments. The same participants will experience greater improved brain activation patterns and an improvement in cognitive functioning compared to placebo controlled subjects.
2. Measure the effects of citicoline on marihuana absorption and metabolism and determine if these changes parallel changes in subjective and physiological responses in a laboratory setting.

   Hypothesis - Chronic (8 weeks) treatment with 2 g/day citicoline will produce increases in subjective and physiological effects of both acute marihuana smoking and placebo marihuana smoking compared to chronic placebo citicoline. Citicoline will have no effect on marihuana pharmacokinetics.
3. Measure the effects of citicoline on marijuana-induced cue-induced craving and brain electrical activity (EEG).

Hypothesis - Chronic (8 weeks) treatment with 2 g/day citicoline will reduce objective measures of marijuana cue-reactivity, and subjective reports of craving in response to marihuana cues will also be attenuated compared to chronic placebo citicoline treatment.

DETAILED DESCRIPTION:
Marijuana dependence is an important public health problem in the United States, yet still no effective therapies are available. It is unclear how marijuana affects brain function after acute or chronic use. Knowing about the changes in brain function during marijuana dependence would aid in the understanding of the neurobiological basis of marijuana abuse and serve as a foundation for the development of new treatment medications for this disorder. New and improved brain imaging techniques, such as functional MRI (fMRI) and magnetic resonance spectroscopy (MRS), allow the viewing of these subtle, yet important, changes in brain function.

Citicoline is used to treat victims of head trauma and neurodegenerative disorders. It has been found to be effective in reducing cocaine use and craving, and it has no known side effects. It has also been shown to reduce marijuana use. This is likely due to citicoline's ability to reduce insomnia and craving, act as a mild antidepressant, and improve cognitive function. How citicoline reduces drug use may be related to effects on cerebral blood flow and/or brain phospholipid metabolism in the reward areas of the brain.

This study will determine whether citicoline alters marijuana use patterns, reduces craving, and affects brain phospholipids and metabolism in marijuana-dependent people. The outcome of the study could offer important insights into the pathophysiology and course of marijuana dependence. Furthermore, this study's outcome could potentially relate to other drug dependence disorders.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current marijuana dependence
* Women with a negative pregnancy test prior to study entry
* Heavy smoker, defined as smoking more than 10 joints per week

Exclusion Criteria:

* Abnormal electrocardiogram (ECG)
* Medical disorder that requires prescription medication
* Psychiatric disorder that requires prescription medication
* Abnormal liver function tests
* Taking herbal preparations
* Taking any over-the-counter medications on a chronic basis
* Pregnancy or breast feeding
* Neurological, infectious, or neoplastic disease
* Currently seeking treatment for marijuana abuse
* Meets criteria for alcohol, cocaine, or opioid dependence

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E. Lukas, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Department of Psychiatry, Belmont, Massachusetts, United States

REFERENCES:
- [Derived] Bracken BK, Penetar DM, Rodolico J, Ryan ET, Lukas SE. Eight weeks of citicoline treatment does not perturb sleep/wake cycles in cocaine-dependent adults. Pharmacol Biochem Behav. 2011 Jun;98(4):518-24. doi: 10.1016/j.pbb.2011.03.003. Epub 2011 Mar 21. PMID 21397626

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Citicoline
Started | 11 | 10
Completed | 9 | 10
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Citicoline | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (7.2) | 27.7 (6.9) | 29.0 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 3 | 5 | 8
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Marijuana Use
Time Frame: Measured for 8 weeks of treatment
Measure: Mean (Standard Error); unit: Reported uses per day
Arm/Group | Placebo | Citicoline
Number analyzed (Participants) | 9 | 10
Reported uses per day | 2.5 (.71) | 3.9 (1.1)

2. Secondary Outcome: Neurocognitive Function
Description: Multiple Source Interference Test (MSIT)
Time Frame: Before and after 8 weeks of treatment
Measure: Mean (Standard Error); unit: Accuracy percent improvement
Arm/Group | Placebo | Citicoline
Number analyzed (Participants) | 9 | 10
Accuracy percent improvement | 32.45 (18.8) | 16.08 (7.9)

ADVERSE EVENTS:
Arm/Group | Placebo | Citicoline
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 1/9 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Citicoline (N=10)
Migraine headache (General disorders) | 1 (1) | 0 (0)
NAusea/Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes